CLINICAL TRIAL: NCT03531216
Title: Psychophysiological Effect of Local Rosemary and Olive Oil Application Onto the Hands of Patients With Systemic Sclerosis - a Prospective Crossover, Open-label, Nonrandomized Trial
Brief Title: Topical Rosemary Oil Application in Systemic Sclerosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ARCIM Institute Academic Research in Complementary and Integrative Medicine (Other)
Collaborators: University Hospital Tuebingen (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ROS_02
Record Dates: First submitted 2018-05-09; First posted 2018-05-21 (Actual); Last update posted 2019-01-10 (Actual); Status verified 2018-05

CONDITIONS: Systemic Sclerosis
MeSH Terms: conditions — Scleroderma, Systemic

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Topical application of rosemary oil (Active Comparator): Rosemary essential oil (10% )
  Interventions: Other: Rosemary essential oil
- Placebo (Placebo Comparator): Pharmaceutical quality olive oil
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Rosemary essential oil — Topically-applied oil to both dorsal and palmar aspects of the hands
  Arms: Topical application of rosemary oil
Other: Placebo — Topically-applied oil to both dorsal and palmar aspects of the hands
  Arms: Placebo

SUMMARY:
The objectives of this prospective crossover, open-label, nonrandomized study are to estimate effect sizes of vasodilatation and sense of warmth after application of topical rosemary essential oil in patients suffering from systemic sclerosis.

DETAILED DESCRIPTION:
In a crossover design, patients suffering from systemic sclerosis (12 subjects) receive applications of olive oil and of 10% Rosmarinus officinalis L. (rosemary) essential oil to both hands with a wash-out period of 3 hours. Effects on vasodilatation are measured with infrared thermography. Patients' sense of warmth is assessed by the "Herdecke warmth perception questionnaire". Measurements take place at baseline and 45 minutes following the interventions (pre-post-comparison). To determine within and between-differences, 2-sample t-tests will be used and effect sizes will be calculated (Standardized Effect Size).

ELIGIBILITY:
Inclusion Criteria:

* Systemic sclerosis with skin involvement of hands and fingers
* Raynaud phenomenon with frequent symptoms of cold hands

Exclusion Criteria:

* Topical treatment with nitroglyceride
* Lymphdrainage < 24 hours
* Other topical treatment of hands and arms < 4 hours prior to study intervention

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2015-11-02 (Actual); Primary Completion 2016-03-21 (Actual); Study Completion 2016-03-21 (Actual)

PRIMARY OUTCOMES:
Change from baseline in temperature at the fingers | baseline and 45 minutes after the intervention
  Distal skin temperature in °C measured at the fingers with a high-definition infrared camera (FLIR-Systems, type SC660) before and 45 minutes following the oil application

SECONDARY OUTCOMES:
Change from baseline in temperature at the back of the hands | baseline and 45 minutes after the intervention
  Distal skin temperature in °C measured at the back of the hands with a high-definition infrared camera (FLIR-Systems, type SC660) before and 45 minutes following the oil application
Change from baseline in temperature at the forearms | baseline and 45 minutes after the intervention
  Distal skin temperature in °C measured at the forearms with a high-definition infrared camera (FLIR-Systems, type SC660) before and 45 minutes following the oil application
Change from baseline of "Herdecke warmth perception questionnaire" (HeWEF) | baseline and 45 minutes after the intervention
  Patients' sense of warmth in different body regions as well as overall warmth assessed before and 45 minutes following the oil application
"Scleroderma Health Assessment Questionnaire" (SHAQ) | baseline
  Questionnaire with 8 sections: e.g. dressing, arising, eating, walking,hygiene, etc... with 2 or 3 questions for each section. Scoring within each section is from0 (without any difficulty) to 3 (unable to do).
Rodnan skin score of the hands | baseline
  Skin score to assess the clinical severity of systemic scleroderma. 17 body areas are assessed by clinical palpation. The examiner assesses the skin thickness using a 4-point scale:0 = normal thickness, 1 = weak skin thickening, 2 = moderate skin thickening, 3 = severe skin thickening.

CONTACTS AND LOCATIONS:
Overall Officials: Jan Vagedes, Dr., Study Director — ARCIM Institute; University of Tuebingen
Locations (2):
- Germany (2):
  - ARCIM Institute, Filderstadt, Baden-Wurttemberg
  - Universitätsklinikum Tuebingen, Abteilung Innere Medizin II, Tübingen, Baden-Wurttemberg